CLINICAL TRIAL: NCT04628689
Title: Comparison Of The Analgesic Efficacy Of Quadratus Lumborum Block By Paraspinous Sagittal Shift Approach With Different Concentrations Of Bupivacaine in Hip Surgeries
Brief Title: Quadratus Lumborum Block by Paraspinous Sagittal Shift Approach With Different Concentrations Of Bupivacaine in Hip Surgeries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, doaa rashwan, Assistant professor Doaa Rashwan, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMBSUREC/01092020/Abd El Badei
Record Dates: First submitted 2020-09-30; First posted 2020-11-13 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Hip Surgeries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 0.25% bupivacaine (Active Comparator): 30 ml 0.25% bupivacaine
  Interventions: Other: quadratus lumborum block by paraspinous sagittal shift approach
- Group 0.375% bupivacaine (Active Comparator): 0.375% bupivacaine
  Interventions: Other: quadratus lumborum block by paraspinous sagittal shift approach

INTERVENTIONS:
Other: quadratus lumborum block by paraspinous sagittal shift approach — quadratus lumborum block by paraspinous sagittal shift approach

SUMMARY:
The aim of this study is to evaluate the optimum concentration of bupivacaine in Paraspinous Sagittal Shift Approach for Quadratus Lumborum Block in hip Surgeries

DETAILED DESCRIPTION:
With the patient in the lateral decubitus and the block side independent, a curvilinear ultrasound transducer (2-5 MHz) will be directed caudally in a sagittal plane 3-4 cm lateral to the lumbar spinous process of L4, which is almost opposite to the iliac crest, producing a longitudinal scan of the lumbar paravertebral region; and thus identifying the transverse processes of L3 and L4, with PM muscle in-between and erector spinae muscle posteriorly.

The probe is shifted slowly to the lateral side until the transverse processes disappear and the QL muscle is evident in its long axis attached caudally to the iliac crest with a characteristic sonographic image of three muscle layers appearing from posterior to anterior as: erector spinae, QL, and PM muscles respectively. After subcutaneous local infiltration with lidocaine at the cephalic end of the probe, the block needle is advanced in a cephalo-caudal direction, through the erector spinae and QL muscles, until it pierces the epimysium of the QL. LA is injected anterior to the QL muscle, observing its spread in a caudal direction towards the iliac crest between the QL and psoas muscles

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II undergoing hip surgery.

Exclusion Criteria:

* Contraindications for regional blocks (eg. Patient refusal Infection at the injection site, coagulopathy) allergic reaction to drugs. opium addiction, any drug or substance abuse

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-11-20 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
time to first request of analgesics | Postoperative 24 hours
  Postoperative time to first request of analgesics (hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Benisuef univercity, Banī Suwayf, Benisuef, Egypt

IPD SHARING:
Plan to Share IPD: No